CLINICAL TRIAL: NCT07331168
Title: EVALUATION OF THE EFFECT OF ACTIVE WARMING APPLIED TO THE MOTHER DURING CESAREAN SECTION ON POST-BREASTFEEDING OUTCOMES: A RANDOMIZED CONTROLLED STUDY
Acronym: ACTIVE WARMING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Bilecik Seyh Edebali Universitesi (Other); Kutahya City Hospital (Other)
Responsible Party: Principal Investigator, Havva Yeşildere Sağlam, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KutahyaHSU_2025
Record Dates: First submitted 2025-11-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Cesarean Resection; Breastfeeding; Thermal Comfort
Keywords: Cesarean; active warming; thermal comfort; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, parallel-group interventional study evaluating the effect of active warming applied to mothers during and after cesarean delivery on early postpartum breastfeeding outcomes. Participants will be randomly assigned, via computer-generated allocation, to either the intervention group receiving active warming or the control group receiving standard care without warming. The study will be conducted in a [single-blind / open-label] manner. The primary objective is to assess the effect of active warming on breastfeeding success, thermal comfort, and perceived insufficient milk supply.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Active warming group
  Interventions: Other: active warming; Other: active warming II
- Control (No Intervention): Control group

INTERVENTIONS:
Other: active warming — During the cesarean section, heating will be applied at 37 degrees. (45 minutes)
  Carbon fiber resistive heating pads are reusable, where a low-voltage electric current flows, causing heat to accumulate in the carbon fibers that make up the blanket's filling. A heating pad will be used to warm participants. This pad has a control unit, is 120 cm long, and is suitable for operating room conditions. It is safe and operates at low voltage. It heats to a maximum of 40 degrees Celsius. In this study, heating will be used to a temperature of 37 degrees Celsius.
  Arms: Intervention
Other: active warming II — After the cesarean section, heating will be applied to the recovery area at 37 degrees. (45 minutes)
  Carbon fiber resistive heating pads are reusable, where a low-voltage electric current flows, causing heat to accumulate in the carbon fibers that make up the blanket's filling. A heating pad will be used to warm participants. This pad has a control unit, is 120 cm long, and is suitable for operating room conditions. It is safe and operates at low voltage. It heats to a maximum of 40 degrees Celsius. In this study, heating will be used to a temperature of 37 degrees Celsius.
  Arms: Intervention

SUMMARY:
Hypothermia is a complication of cesarean section and a cause of breastfeeding problems. Preventing maternal hypothermia is one of the goals of the enhanced postoperative recovery (ERAS) protocol and is important for the health of both mother and baby. This clinical trial aims to determine the effects of active warming during and after cesarean delivery on breastfeeding outcomes, thermal comfort, and perceived insufficient milk supply.

The primary questions it aims to answer are:

1. To evaluate the effect of active warming during cesarean delivery on mothers' perception of thermal comfort.
2. To evaluate the effect of active warming after cesarean delivery on mothers' perceived insufficient milk supply.
3. To determine the effect of active warming after cesarean delivery on breastfeeding success.

Participants:

Warming will be provided using an active warming bed during cesarean delivery (45 minutes). Warming will continue in the postpartum care unit (45 minutes).

The control group will not receive any warming and will receive the hospital's standard care procedure.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Primiparous, singleton pregnancy
* Gestational age >37 weeks, elective cesarean section under spinal anesthesia
* No issues with breastfeeding the baby or herself during the postpartum period
* Voluntarily participating

Exclusion Criteria:

* Those with a gestational age of less than 37 weeks,
* Those with an urgent delivery decision or those with accompanying comorbidities (severe preeclampsia, placenta previa, placental abruption, umbilical cord prolapse, fetal distress),
* those with multiple pregnancies,
* those with a core body temperature above 37.5 °C,
* those who started cesarean delivery with spinal anesthesia and later switched to general anesthesia due to complications,
* those with known impaired thermoregulation or thyroid disorder

Translated with DeepL.com (free version)

-

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Success | Postperative Day 1- First breastfeeding session
  Evaluation will be performed using the LATCH breastfeeding diagnostic tool. The LATCH Breastfeeding Assessment Scale consists of 5 sub-dimensions: Latch, Audible swallowing, Type of nipple, Comfort, and Hold.
  Each item is scored between 0 and 2 points. The total score ranges from 0 to 10. Higher scores indicate more effective and successful breastfeeding.
Breastfeeding success | Postoperative Day 1, 24.hour
  Evaluation will be performed using the LATCH breastfeeding diagnostic tool. The LATCH Breastfeeding Assessment Scale consists of 5 sub-dimensions: Latch, Audible swallowing, Type of nipple, Comfort, and Hold.
  Each item is scored between 0 and 2 points. The total score ranges from 0 to 10. Higher scores indicate more effective and successful breastfeeding.
Perception of insufficient milk | Postoperative Day 1, First breastfeeding session
  Assessment will be made using the Insufficient Milk Perception Scale. The Perception of Insufficient Milk (PIM) Scale is used to assess mothers' subjective perceptions of whether their milk supply is sufficient to feed their infants. The scale consists of items that question the mother's perception of milk quantity, infant satisfaction, and the adequacy of breastfeeding. Items are generally scored using a Likert scale, and the total score ranges between predetermined minimum and maximum values. Higher scores indicate a higher level of perceived insufficiency in the mother's milk supply. A score of "0" indicates that milk is perceived as completely insufficient, while a score of "10" indicates that milk is perceived as completely sufficient. The scale is scored from 0 to 50. A higher score indicates a higher perception of milk sufficiency.
Perception of insufficient milk | Postoperative Day 1, 24. hour
  The assessment will be performed using the Insufficient Milk Perception Scale. The Perception of Insufficient Milk (PIM) Scale is used to assess mothers' subjective perceptions of whether their milk supply is sufficient to feed their infants. The scale consists of items that question the mother's perception of milk quantity, infant satisfaction, and the adequacy of breastfeeding. Items are generally scored using a Likert scale, and the total score ranges between predetermined minimum and maximum values. Higher scores indicate a higher level of perceived insufficiency in the mother's milk supply. A score of "0" indicates that milk is perceived as completely insufficient, while a score of "10" indicates that milk is perceived as completely sufficient. The scale is scored from 0 to 50. A higher score indicates a higher perception of milk sufficiency.
Thermal comfort | Preoperative Day 1, Before the cesarean section
  The Thermal Comfort Perception Scale will be used. The Thermal Comfort Scale is a subjective scale used to assess how comfortable, acceptable, or uncomfortable individuals perceive the temperature conditions of their environment. The scale is generally a single-item or multi-item structure that questions the perception of hot-cold and the level of thermal comfort. Scores range between predetermined minimum and maximum values, with higher scores indicating a higher level of thermal comfort and lower scores indicating thermal discomfort. The scale is a 5-point Likert type with options of 1 "none", 2 "somewhat", 3 "moderately", 4 "a lot", and 5 "very much". The lowest possible score on the 11-item scale is 11, and the highest is 49.
Thermal comfort II | Day 1, During the cesarean section (at 15 minutes)
  The Temperature Comfort Perception Scale will be used. The Thermal Comfort Perception Scale will be used. The Thermal Comfort Scale is a subjective scale used to assess how comfortable, acceptable, or uncomfortable individuals perceive the temperature conditions of their environment. The scale is generally a single-item or multi-item structure that questions the perception of hot-cold and the level of thermal comfort. Scores range between predetermined minimum and maximum values, with higher scores indicating a higher level of thermal comfort and lower scores indicating thermal discomfort. The scale is a 5-point Likert type with options of 1 "none", 2 "somewhat", 3 "moderately", 4 "a lot", and 5 "very much". The lowest possible score on the 11-item scale is 11, and the highest is 49.
Thermal comfort III | Postoperative Day 1,After the cesarean section (at 30 minutes)
  The Thermal Comfort Perception Scale will be used. The Thermal Comfort Scale is a subjective scale used to assess how comfortable, acceptable, or uncomfortable individuals perceive the temperature conditions of their environment. The scale is generally a single-item or multi-item structure that questions the perception of hot-cold and the level of thermal comfort. Scores range between predetermined minimum and maximum values, with higher scores indicating a higher level of thermal comfort and lower scores indicating thermal discomfort. The scale is a 5-point Likert type with options of 1 "none", 2 "somewhat", 3 "moderately", 4 "a lot", and 5 "very much". The lowest possible score on the 11-item scale is 11, and the highest is 49.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It may be shared if contacted by the researcher for reasonable reasons.

REFERENCES:
- [Background] Zhuo Q, Xu JB, Zhang J, Ji B. Effect of active and passive warming on preventing hypothermia and shivering during cesarean delivery: a systematic review and meta-analysis of randomized controlled trials. BMC Pregnancy Childbirth. 2022 Sep 21;22(1):720. doi: 10.1186/s12884-022-05054-7. PMID 36131231
- [Background] Yigit F, Cigdem Z, Temizsoy E, Cingi ME, Korel O, Yildirim E, Ovali F. Does warming the breasts affect the amount of breastmilk production? Breastfeed Med. 2012 Dec;7(6):487-8. doi: 10.1089/bfm.2011.0142. Epub 2012 Mar 16. PMID 22424466
- [Background] Talhaoglu D, Baser M, Ozgun MT. The Effects of Actively Warming the Patient on Maternal and Infant Well-Being in a Cesarean Section Operation. J Perianesth Nurs. 2024 Jun;39(3):366-374. doi: 10.1016/j.jopan.2023.08.008. Epub 2024 Jan 12. PMID 38219080
- [Background] Ozkan H, Uzun Ozer B, Ari O. The Effect of Hot Application Applied to the Breast with the Help of the Thera Pearl in the Postpartum Period on Mothers' Milk Perception and Postpartum Breastfeeding Self-Efficacy: A Randomized Controlled Study. Healthcare (Basel). 2024 May 8;12(10):968. doi: 10.3390/healthcare12100968. PMID 38786381
- [Background] Kholeif MFMA, Herpertz GU, Brauer A, Radke OC. Prewarming Parturients for Cesarean Section Does Not Raise Wound Temperature But Body Heat and Level of Comfort: A Randomized Trial. J Perianesth Nurs. 2024 Feb;39(1):58-65. doi: 10.1016/j.jopan.2023.06.001. Epub 2023 Sep 9. PMID 37690018
- [Background] Duryea EL, Nelson DB, Wyckoff MH, Grant EN, Tao W, Sadana N, Chalak LF, McIntire DD, Leveno KJ. The impact of ambient operating room temperature on neonatal and maternal hypothermia and associated morbidities: a randomized controlled trial. Am J Obstet Gynecol. 2016 Apr;214(4):505.e1-505.e7. doi: 10.1016/j.ajog.2016.01.190. Epub 2016 Feb 10. PMID 26874298
- [Background] Alshakhs FH, Katooa NE, Badr HA, Thabet HA. The Effect of Alternating Application of Cold and Hot Compresses on Reduction of Breast Engorgement Among Lactating Mothers. Cureus. 2024 Jan 28;16(1):e53134. doi: 10.7759/cureus.53134. eCollection 2024 Jan. PMID 38420104